CLINICAL TRIAL: NCT05250895
Title: Molecular Imaging of the Hypoxic Tumor Microenvironment to Predict Response to Yttirum-90 Selective Internal Radiation Therapy in Hepatocellular Carcinoma- Pilot Study
Brief Title: BOLD MRI and FMISO PET for the Assessment of Hypoxic Tumor Microenvironment in Patients with Oligometastatic Liver Cancer Undergoing Yttirum-90 Selective Internal Radiation Therapy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Brandon, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00002804; NCI-2021-09943 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00002804; RAD5342-21 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2021-12-22; First posted 2022-02-22 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: BCLC Stage a Hepatocellular Carcinoma; BCLC Stage B Hepatocellular Carcinoma; BCLC Stage C Hepatocellular Carcinoma; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — fluoromisonidazole; Biopsy; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (18F-fluoromisonidazole, PET, DCE MRI) (Experimental): Patients receive 18F-fluoromisonidazole IV and undergo PET and DCE MRI within 30 days before beginning Y90 SIRT. Patients undergo Y90 SIRT per standard of care.
  Interventions: Other: 18F-Fluoromisonidazole; Procedure: Biopsy; Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Other: 18F-Fluoromisonidazole — Given IV
  Other Names: 18F-MISO; 18F-Misonidazole; FMISO
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging — Undergo DCE MRI
  Other Names: DCE; DCE MRI; DCE-MRI; DYNAMIC CONTRAST ENHANCED MRI
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This early phase I trial evaluates the use of hypoxia (lack of oxygen) as a measure in determining the outcome of Y90 selective internal radiation therapy in patients with liver cancer that has spread to a limited number of sites (oligometastatic). Radioembolization with Y90 is a minimally invasive procedure that combines embolization and radiation therapy to treat metastatic liver cancer. Tiny beads filled with radioactive isotope Y-90 are placed inside the blood vessel that provide blood supply to the tumor. This will block the blood flow to the tumor cells while providing a high radiation dose without harming healthy normal tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To investigate the variability of hypoxia in hepatocellular carcinoma (HCC) as quantified by blood oxygen level-dependent (BOLD) magnetic resonance imaging (MRI) and dynamic 18F-Fluoromisonidazole (FMISO) positron emission tomography (PET).

SECONDARY OBJECTIVES:

I. Investigate whether hypoxia, as quantified by BOLD MRI, dynamic FMISO PET, HIF-1alpha and VEGF expression, predicts HCC response to yttrium-90 (Y90) selective internal radiation therapy (SIRT).

II. Assess whether hypoxia quantification by BOLD MRI, dynamic FMISO, HIF-1alpha or VEGF expression individually or in combination more accurately predict the degree of HCC tumor response to Y90 SIRT.

III. Compare the tumor dose response threshold between hypoxic and non-hypoxic HCCs treated with Y90 SIRT.

OUTLINE:

Patients receive 18F-fluoromisonidazole intravenously (IV) and undergo PET and dynamic contrast enhanced (DCE) MRI within 30 days before beginning Y90 SIRT. Patients undergo Y90 SIRT per standard of care.

After completion of study intervention, patients are followed up at 90 days, and then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Established HCC diagnosis, unilobar or bilobar disease
* At least 1 tumor >= 3 cm
* Oligometastatic disease
* Barcelona Clinic Liver Cancer (BCLC) stage A, B or C
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy > 12 weeks as determined by the Investigator
* The effects of Y90 Radioembolization on the developing human fetus are unknown. For this reason, female of child-bearing potential (FCBP) must have a negative serum or urine pregnancy test prior to starting therapy
* FCBP and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* A female of childbearing potential (FCBP) is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months

Exclusion Criteria:

* Patients who are definite transplant candidates
* Concurrent second malignancy outside of the liver
* Infiltrative liver tumor
* Previous liver-directed therapy to targeted tumors
* BCLC stage D
* Bilirubin > 2 mg/dL for lobar treatment and bilirubin > 3 mg/dL for segmental or bi-segmental Y90-SIRT
* Albumin < 3 g/dL
* Projected lung dose of > 30 Gy in a single session to the liver after prospective treatment planning
* Body mass index (BMI) > 40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
To investigate the variability of hypoxia in HCC at baseline as quantified by BOLD MRI | From weeks 1-2 up to 1 year
  Threshold <1.0 R2 tumor to normal ratio (no unit) as a cutoff for hypoxia
To investigate the variability of hypoxia in HCC at baseline as quantified by immunohistochemistry | From weeks 1-2 up to 1 year
  The staining intensity will be measured and scored with four scales: no staining=0, weak staining=1, moderate staining=2, and strong staining=3. The final staining score will be obtained by stained stumor area% x positive tumor cells % x staining intensity. The tumors will be then categorized as hypoxic (scores 8 to 16) vs. non-hypoxic (scores 0 to 7) (no units).

SECONDARY OUTCOMES:
Determine whether hypoxia is predictor of response in HCC treated with Y90 SIRT | From week 0 up to 1 year
  Treatment Response Assessment using mRECIST
Treatment response | From week 0 Up to 1 year
  Assessed using modified Response Evaluation Criteria in Solid Tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Nima Kokabi, MD, FRCPC, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States